CLINICAL TRIAL: NCT01627925
Title: Safety Study of Positive Airway Pressure Via a Nasal Mask on Upper Airway Patency During Induction of Anesthesia in Obese Patients
Brief Title: Safety Study of Positive Airway Pressure Via a Nasal Mask in Obese Patients
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Responsible Party: Principal Investigator, Yandong Jiang, associated professor, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2012-P-000054
Record Dates: First submitted 2012-06-22; First posted 2012-06-26 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Upper Airway Obstruction
Keywords: nasal positive airway pressure; upper airway obstruction; mask ventilation
MeSH Terms: conditions — Airway Obstruction | interventions — Continuous Positive Airway Pressure

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Face mask and nasal mask without PEEP (Experimental): Face mask ventilation and nasal mask ventilation without PEEP
  Interventions: Device: nasal mask and continuous positive airway pressure
- Nasal mask and face mask with PEEP (Experimental): Nasal mask ventilation and face mask ventilation with PEEP
  Interventions: Device: nasal mask and continuous positive airway pressure

INTERVENTIONS:
Device: nasal mask and continuous positive airway pressure — nasal mask use instead of face mask application of continuous positive airway pressure during induction of general anesthesia
  Other Names: nasal mask (Contour delux, Respironics)

SUMMARY:
Upper airway obstruction (UAO) is a frequently occurring complication during induction of general anesthesia. The American Society of Anesthesiologist (ASA) closed claim analysis of anesthesia complications indicate that a difficult airway is one of the most challenging scenarios continuously facing anesthesia providers.

The mechanism of UAO during anesthesia has not been well understood. Posterior displacement of soft palate, tongue and epiglottis are believed to be the primary contributing factors. Obesity is well known to be an essential characteristic which reflects propensity to UAO. The mechanism of UAO during anesthesia shares many similarities with the upper airway obstruction observed during obstructive sleep apnea (OSA). Nasal continuous positive airway pressure (nCPAP) via nasal mask (NM) can maintain the airway patent with near 100% success in patients with OSA. Obesity is a major risk factors for obstructive sleep apnea and obese patients have a higher prevalence of UAO during anesthesia. Therefore, the investigators hypotheses that nCPAP should eliminate airway obstruction in obese patients under anesthesia. The investigators propose to test this hypothesis and determine the efficacy of nCPAP on maintaining airway patency in obese patients who require general anesthesia.

DETAILED DESCRIPTION:
Upper airway obstruction (UAO) is an unpredictable and frequently occurring complication during induction of general anesthesia. Since obese patients ( BMI>30 km/ m2) are more vulnerable to develop airway obstruction either during sleep or under anesthesia, and the segment of obese individuals in the entire population keep growing, difficult airway management under anesthesia becomes even more challenging than ever. The most serious event related to difficult airway management under anesthesia is "cannot intubate, cannot ventilate". Unfortunately, even with modern technologic advances, 16% of death and permanent brain damage related to anesthesia have been attributed to failure of difficult airway management 3. The American Society of Anesthesiologist (ASA) closed claim analysis of anesthesia complications indicate that a difficult airway is one of the most challenging scenarios continuously facing anesthesia providers. Indeed, it can be a fatal complication of general anesthesia. Therefore, measures used to reduce the incidence of difficult airways during anesthesia remain to be improved.

The mechanism of UAO during anesthesia has not been well understood. Posterior displacement of soft palate, tongue and epiglottis are believed to be the primary contributing factors. Obesity is well known to be an essential characteristic which reflects propensity to UAO. Accordingly, obese patients are a high-risk group for perioperative airway catastrophe and prone to develop progressively narrower pharyngeal airways due to an increase of soft tissue volume surrounding the pharyngeal airway. More and more evidence indicates that the mechanism of UAO during anesthesia shares many similarities with the upper airway obstruction observed during obstructive sleep apnea (OSA). Nasal continuous positive airway pressure (nCPAP) via nasal mask (NM) can maintain the airway patent with near 100% success in patients with OSA, if they can tolerate it. Under anesthesia, tolerance should not be an issue as the patient is anesthetized. Obesity is a major risk factors for obstructive sleep apnea and obese patients have a higher prevalence of UAO during anesthesia. Therefore, the investigators hypotheses that nCPAP should eliminate airway obstruction in obese patients under anesthesia. The investigators propose to test this hypothesis and determine the efficacy of nCPAP on maintaining airway patency in obese patients who require general anesthesia.

ELIGIBILITY:
Inclusion Criteria:

* Thirty-two subjects with BMI limited in the range of 30 km/ m2 to 50 km/m2 and age of 18-65 years will be enrolled. Subjects must also meet ASA physical status classification I-III, require general anesthesia for elective surgery and be able to breathe through both their nose and mouth while awake.

Exclusion Criteria:

* 1. Patients with major cardiovascular disease, respiratory disease, cerebral vascular disease or American Society of Anesthesiologists physical status class IV or greater.

  2. Abnormal vital signs on the day of admission for surgery [heart rate (HR, >100 bpm or <40 bpm), blood pressure (BP, >180/100 mmHg or <90/60 mmHg), room air transcutaneous oxyhemoglobin saturation (SPO2) <96%] that are not correctable with his or her routine medication or commonly used pre-operative medication.

  3. Having claustrophobia and not able to tolerate the mask. 4. Any person with an anticipated difficult airway or those with a history of difficult airway. This will include subjects who require or may require either a fiberoptic intubation or intubation while awake.

  5. Gastric-esophageal reflex disease that is refractory to treatment or a full stomach.

  6. The subject has been in bed for more than 24 hours. 7. Neurological symptoms associated with neck extension, a neurological deficit from a previous stroke or spinal cord injury, a recent stroke or transient ischemic attack (TIA) within 2 weeks.

  8. Pregnant women and women less than one month post-partum. Ruling out pregnancy will be conducted by careful history and physical examination as performed routinely prior to surgery. If the history is believed to be unreliable, the patient will be excluded unless a pregnancy test is performed and the result of the test is negative.

  9. Emergency cases and subjects who have not adhered to the ASA NPO (Nil Per Os) guidelines.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-06; Primary Completion 2013-04 (Estimated); Study Completion 2013-06 (Estimated)

PRIMARY OUTCOMES:
Expired tidal volume | About two minute during induction of general anesthesia

SECONDARY OUTCOMES:
Volume of CO2 | About two minute during induction of general anesthesia

CONTACTS AND LOCATIONS:
Overall Officials: Yandong Jiang, MD, PhD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States